CLINICAL TRIAL: NCT02419365
Title: International Prospective Primary Ciliary Dyskinesia (PCD) Registry for Systematic Data Collection on Incidence, Clinical Presentation, Treatment and Course of the Disease
Brief Title: International Primary Ciliary Dyskinesia (PCD) Registry
Acronym: PCDregistry
Status: Recruiting | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: European Commission (Other); University of Nicosia (Other); Rigshospitalet, Denmark (Other); KU Leuven (Other); Hannover Medical School (Other); Attikon Hospital (Other); Amsterdam UMC, location VUmc (Other); University of Bern (Other); University of Southampton (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); University of North Carolina (Other); Ruhr University of Bochum (Other); Federico II University (Other); Hospital Vall d'Hebron (Other); Medical University of Vienna (Other); Marmara University (Other); University Hospital, Martin (Other); University of Pisa (Other); Assistance Publique - Hôpitaux de Paris (Other); University of Alberta (Other); University of Giessen (Other)
Responsible Party: Principal Investigator, Petra Pennekamp, Dr, University Hospital Muenster
Other Study IDs: PCD Registry
Record Dates: First submitted 2014-02-03; First posted 2015-04-17 (Estimated); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Primary Ciliary Dyskinesia (PCD)
Keywords: Primary Ciliary Dyskinesia (PCD)
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PCD: Individuals with Primary Ciliary Dyskinesia will be assessed in a pure observational design without intervention

SUMMARY:
The purpose of the international prospective PCD Patient Registry is to systematically measure, survey and compare different aspects of PCD manifestation, course and treatment, to provide data for epidemiological research and to identify special patient groups suitable for multi-center trials.

This International PCD Registry is also part of the European Reference Network ERN-LUNG. We follow the recommendations of the EU Expert Committee on Rare Diseases (EUCERD), which recommend an international interoperability of registries and databases to pool and exchange knowledge and data on rare diseases.

DETAILED DESCRIPTION:
PCD is a rare disorder of mucociliary clearance caused by defective hair like organelles (cilia). The purpose of the PCD Registry is to measure, survey and compare different aspects of PCD manifestation, course and treatment, to provide data for epidemiological research and to identify special patient groups suitable for multi-centre trials.

The PCD Registry is part of the European Reference Network for Rare Lung Diseases ERN-LUNG (https://ern-lung.eu/). We follow the recommendations of the EU Expert Committee on Rare Diseases (EUCERD), which recommend an international interoperability of registries and databases to pool and exchange knowledge and data on rare diseases.

How can the data be entered to the registry? The data can either be entered into the PCD Registry directly after login, or imported via a specific *CSV file that we provide in advance (download option after Log In or e-mail request to PCDregistry.eu@ukmuenster.de, Simone.Helms@ukmuenster.de or Petra.Pennekamp@ukmuenster.de).

Under special circumstances (e.g. import of existing datasets from other registries/cohorts) we provide support to enter your data. The PCD Registry is accessible from the web. Each authorised operator is able to enter the data for their country/centre and export own center specific data to different formats (CSV/Microsoft Excel, PDF, SAS, Stata, R, ODM or SPSS).

A highly protected system will ensure data protection through the encryption of data. Identifying patient data are not collected in the PCD Registry.

Where are the data stored? At the University of Muenster, Institute of Medical Informatics - Informatics for personalised medicine (IMI). A server is located in secure premises, where access is allowed to authorized personnel only. Data storage is in agreement with EU data protection legislation.

How to become a PCD Registry Centre? In order to get assigned as a referring centre please contact the administration under PCDregistry.eu@ukmuenster.de, Simone.Helms@ukmuenster.de and Petra.Pennekamp@ukmuenster.de.

Information for PCD Patients:

Why do we need a PCD Registry? Registries are the only way to pool data in the field of Rare Diseases (RD) such as PCD in order to achieve a sufficient sample size for epidemiological and/or clinical research. RD Registries such as the PCD Registry constitute key instruments to develop clinical research in the field of RD, to improve patient care and healthcare planning. RD Registries such as the PCD Registry are vital to assess the feasibility of clinical trials, to facilitate the planning of appropriate clinical trials and to support the enrolment of patients.

Why should I as a patient participate? Patient involvement is the key factor in the establishment of any patient registry, especially RD Registries. For the purpose of the above aims, we need as many patients in the PCD Registry as possible in order to make sure that data are representative of the whole spectrum of the disease and to have enough patients to render research possible - research that may benefit you or other patients in the future.

I you - as a patient - have further questions please do not hesitate to contact us.

Which data are collected? We collect demographic data (e.g. current age, sex, age, diagnostic findings and symptoms at diagnosis) but also clinical data which are recorded (e.g. lung function, weight, height, infections, treatment and complications). The data are collected using a common set of definitions, following the recommendations of the EU Expert Committee on Rare Diseases (EUCERD). This ensured international interoperability of registries and databases to pool and exchange knowledge and data on rare diseases.

Ways to register:

Registration will be performed by the treating physician via password-secured access. The access authorization, as well as the necessary password will be passed on by the PCD Registry administrator (Simone.Helms@ukmuenster.de).

Information about data security:

To ensure that patients are not accidentally registered twice and to take into account a changing of caring physician, personal data such as month and year of birth have to be included in the first step of patient registration. These will be directly transferred into a Patient identification-Code (PID) and automatically generated pseudonym. Tracking a patient's identification with the PID is impossible. Other identifying data such name, initials or day of birth will not be nor recorded. Data saving underlies the regulations for data security laws and the medical confidentiality. International regulations for good clinical practice (GCP) always apply. Unauthorized third parties will not have access to registry data.

Inclusion criteria:

The PCD Patient Registry is a longitudinal study. It recruits all prevalent subjects with PCD and all subsequent incident cases. Patients who fulfil the diagnostic criteria below should be included in the registry

* Clinical presentation consistent with PCD and
* Confirmation of the diagnose by at least two of the following methods
* abnormally low nasal NO concentration/production
* abnormal high frequency video microscopic (HVMA) finding
* abnormal immunofluorescence (IF) finding
* demonstration of biallelic disease-causing mutations by genotyping (Note: in those cases, where genetic diagnosis is not possible because of financial or structural issues, genetic diagnosis can be offered in the framework of a research project)
* abnormal transmission electron microscopy (TEM) finding (Note: if only high frequency video microscopy and nasal NO concentration/production are abnormal, high frequency video microscopy should be repeated at least three times and show the same abnormal results each time)

Given the complexity of diagnosing PCD, not all patients will meet the above mentioned definite diagnostic criteria. Therefore, individuals with typical clinical symptoms and only one abnormal diagnostic test are also eligible to enter the registry.

Ethics and Patient Confidentiality:

Obtaining the necessary patient consents is a prerequisite for entering data in the PCD Registry. As legislation differs in each participating country, it is important to check the requirements with your local Data Protection Officers and Ethics Committees. If you have any questions, please contact PCDregistry.eu@ukmuenster.de or Simone.Helms@ukmuenster.de. You will get support for the Ethics Committee approval procedure, e.g. sample consent forms for Patient Information and Consent. Patients can only be entered into the PCD Registry once you have received their signed, informed consent to do so. Please store all the consent forms that your patients have signed safely at your local institution. It is the responsibility of the reporting centres/countries/registries to have the acquired permissions to export/report data to the PCD Registry.

Data Security:

Due to data protection regulations, the data stored in the server of the PCD Registry must be anonymous (i.e. the patient must not be identifiable). Therefore, the authorised operator has to keep a logbook with the identifying patient data and the code generated by the registry software. It is your responsibility to make sure that access to this list of names and matching patient codes is restricted to authorized personnel only. Furthermore, please note that if your list of matching codes and full names is lost, it will be impossible to retrieve the data identification by means of the PCD Registry software. Moreover, data are encrypted (i.e. not de-codable) when transmitted. The PCD Registry is protected according to EU Data Protection legislation, both physically and technically, and backup is secured.

Funding:

The establishment of the PCD Registry was part of the EU funded BESTCILIA project (FP7 2007-2013) under grant agreement no 305404 (BESTCILIA). Funding continues within several projects including REGISTRY WAREHOUSE (HORIZON2020, GA no 777295)

About us:

The PCD Registry has been designed and established by the BESTCILIA consortium headed by Heymut Omran, University Children's Hospital Muenster, Department of General Pediatrics, Muenster, Germany and is part of the European Reference Network on Rare Lung Diseases ERN-LUNG. For more information, please contact PCDregistry.eu@ukmuenster.de Simone.Helms@ukmuenster.de, Petra.Pennekamp@ukmuenster.de or Johanna.Raidt@ukmuenster.de

ELIGIBILITY:
Inclusion Criteria

Patients of any age who fulfil the diagnostic criteria below are eligible:

Clinical presentation consistent with PCD and consistent findings specific for PCD in at least two of the following methods:

high frequency video microscopic finding transmission electron microscopy finding immunofluorescence finding low nasal NO concentration/production demonstration of biallelic disease-causing mutations by genotyping

Given the complexity of diagnosing PCD, it is anticipated that not all patients will meet these definite diagnostic criteria. Therefore, individuals with typical clinical symptoms and only one abnormal diagnostic test are also eligible to enter the registry. These cases usually are considered to have a possible PCD diagnosis with exceptions made on an individual basis.

Exclusion Criteria Failure or unwillingness to give written informed consent. Missing qualification to perform legal acts or insufficient cognitive ability to give informed consent. A second disease is no exclusion criteria for including data in the PCD-Registry, especially since it is one of the fundamental goals, to learn about co-morbidities.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a diagnosis of Primary Ciliary Dyskinesia.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-01; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
descriptive analysis | 10 years
  Descriptive statistical methods, i.e. frequency tables, location and scale statistics and graphical presentations will be applied to analyse: age at diagnosis, family history (consanguinity), associated malformations/diseases, laterality defects, clinical manifestations (otitis media, rhinosinusitis, pneumonia, bronchiectasis, neonatal respiratory distress syndrome), microbiological results, diagnostic findings (video microscopy, electron microscopy, nasal NO, immunofluorescence analysis), lung function, radiological findings and therapeutic measures (inhalation therapy, antibiotics, oxygen, ventilation, upper airways surgery, lung surgery). Furthermore, quality of life will be assessed using QOL-PCD, a disease specific questionnaire.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Münster, Münster, North Rhine-Westphalia
  - University Hospital Muenster, Department of General Pediatrics, Münster

REFERENCES:
- [Derived] Werner C, Lablans M, Ataian M, Raidt J, Wallmeier J, Grosse-Onnebrink J, Kuehni CE, Haarman EG, Leigh MW, Quittner AL, Lucas JS, Hogg C, Witt M, Priftis KN, Yiallouros P, Nielsen KG, Santamaria F, Uckert F, Omran H. An international registry for primary ciliary dyskinesia. Eur Respir J. 2016 Mar;47(3):849-59. doi: 10.1183/13993003.00776-2015. Epub 2015 Dec 8. PMID 26659107
- See also: ERN-LUNG is a patient-centric network of European healthcare providers and patient organisations, committed Europe-wide and globally to reducing morbidity and mortality from rare lung diseases in people of all ages — https://ern-lung.eu/
- See also: European Platform on Rare Disease Registration — https://eu-rd-platform.jrc.ec.europa.eu/